CLINICAL TRIAL: NCT06059664
Title: The EFfect of FinErenone in Kidney TransplantiOn Recipients: The EFFEKTOR Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-1867
Record Dates: First submitted 2023-08-22; First posted 2023-09-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; Complications
Keywords: Finerenone; Cardiovascular Outcomes; Albuminuria; eGFR decline; Congestive Heart Failure; Kidney biopsy; Functional MRI
MeSH Terms: conditions — Albuminuria; Heart Failure | interventions — finerenone; Sugars

STUDY DESIGN:
Intervention Model Description: 150 kidney transplant recipients will be randomized in a 2:1 ratio to finerenone versus placebo, with an embedded biopsy substudy in 50 participants (25 finerenone/25 placebo) who undergo a research kidney biopsy prior to randomization and at the end of active treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Finerenone (Experimental): Participants in this study arm will receive the study drug Finerenone.
  Initial Dosing: Dosing regimen of 10 mg or 20 mg once daily (QD), based upon screening eGFR. For eGFR < 60 mL/min/1.73m^2, participants will start at 10 mg QD. For eGFR ≥ 60 mL/min/1.73m^2, participants will start at 20 mg QD.
  Dose Titration: Dose will be titrated according to potassium levels. For participants initiated at 10mg, the dose will be up titrated to 20 mg if the potassium level measured after 2 weeks is ≤4.8 meq/L and eGFR has not decreased by >30 percent of the screening visit value. Study drug dosing may be titrated up or down per the below.
  Potassium level: ≤ 4.8
  * If on lower dose, up-titrate to higher dose
  * If on higher dose, continue on the same dose
  Potassium level: 4.9-5.5 = continue same dose
  Potassium level: >5.5 = withhold study drug and recheck potassium within 3 days. Re-initiate study drug at the 10 mg dose once potassium is ≤4.8 meq/L.
  Interventions: Drug: Finerenone Oral Tablet
- Placebo (Placebo Comparator): Participants in this study arm will receive the placebo comparator.
  Initial Dosing: Dosing regimen of 10 mg or 20 mg once daily (QD), based upon screening eGFR. For eGFR < 60 ml/min/1.73m^2, participants will start at 10mg QD. For eGFR ≥ 60ml/min/1.73m^2, participants will start at 20 mg QD.
  Dose Titration: Dose will be titrated according to potassium levels. For participants initiated at 10 mg, the dose will be up titrated to 20 mg if the potassium level measured after 2 weeks is ≤4.8 meq/L and eGFR has not decreased by >30 percent of the screening visit value. Study drug dosing may be titrated up or down per the table below.
  Potassium level: ≤ 4.8
  * If on lower dose, up-titrate to higher dose
  * If on higher dose, continue on the same dose
  Potassium level: 4.9-5.5 = continue same dose
  Potassium level: >5.5 = withhold study drug and recheck potassium within 3 days. Re-initiate study drug at the 10 mg dose once potassium is ≤4.8 meq/L.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone Oral Tablet — Blinded study of finerenone vs. placebo in kidney transplant recipients. Participants will take finerenone or placebo once daily for 12 months. The drug will be up- or down-titrated according to potassium levels.
  Other Names: Kerendia
  Arms: Finerenone
Drug: Placebo — Blinded study of finerenone vs. placebo in kidney transplant recipients. Participants will take finerenone or placebo once daily for 12 months. The drug will be up- or down-titrated according to potassium levels.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
EFFEKTOR is a vanguard, multicenter, phase 2 randomized, double blinded, placebo controlled clinical trial to determine the feasibility, tolerability, safety, and efficacy of finerenone in kidney transplant recipients (KTRs). One hundred fifty (150) KTRs will be randomized in a 2:1 ratio of finerenone to placebo, with two embedded substudies: (i) a kidney biopsy substudy in 50 participants who undergo a research kidney biopsy prior to randomization and at the end of active treatment; and (ii) a functional MRI (fMRI) substudy in 50 participants who undergo fMRI prior to randomization and at the end of active treatment.

DETAILED DESCRIPTION:
Kidney transplantation yields significant improvements in morbidity, mortality, and quality of life for patients with end-stage kidney disease (ESKD), however, the burden from progressive chronic kidney disease (CKD), cardiovascular (CV) events and death remain high. CKD is the result of several pathologic processes, including diabetic and hypertensive sclerosis, calcineurin inhibitor toxicity (CNIT), chronic inflammation and fibrosis that ensues post-acute rejection episodes and other nonspecific insults that can result in CKD mediators. Currently, mean allograft survival is currently 8 years and 12 years for deceased and living donor kidney transplants, respectively. More than 80% of KTRs are under 65 years and 60% under age 55 years, indicating most KTRs will either require a second transplant or eventually transition to maintenance dialysis which portends a poor prognosis and decreased quality of life. CV disease is also highly prevalent, with KTRs having 50 times the annual rate of fatal or nonfatal cardiovascular events and up to 10 times the rate of cardiac death as the general population. Specifically, heart failure is common, with 19% of KTRs sustaining a new diagnosis of heart failure just 3 years post-transplant, and a mean 5.7-7.1 Congestive heart failure (CHF) acute care utilization episodes per 100 person-years. Moreover, kidney and cardiovascular health are tightly intertwined, with kidney disease inciting and exacerbating cardiovascular pathology and vice versa. Thus, there is a critical need for improvements in post kidney transplantation cardiovascular morbidity, mortality, and allograft survival.

Finerenone, a potent, selective, nonsteroidal mineralocorticoid receptor antagonist (MRA), has been shown to significantly reduce the risk of incident worsening CKD and ESKD, as well as preventing major adverse CV events and death in persons with diabetes and native CKD. The pathogenetic mechanisms through which finerenone acts are incompletely understood, but involve reduction of inflammation and fibrosis, key factors in the pathogenesis of CKD and CV disease in KTRs. Moreover, there are preliminary data to suggest that any renin-angiotensin aldosterone system (RAAS blockade), but particularly MRAs and finerenone, could be important to mitigating the effects of CNIT, a significant contributor to graft loss. While current, published clinical trials have been in people with type 2 diabetes and CKD, there is compelling evidence to suggest that these benefits will extend to people with CKD in the absence of diabetes.

Given the high cardiovascular and kidney disease burden in KTRs, and compelling evidence for finerenone in kidney and cardiac protection in patients with native CKD, a vanguard clinical trial of finerenone in 150 KTRs will be undertaken using a randomized, double blind, placebo-controlled study design over the course of 13 months.

Objective 1: To determine the feasibility of recruitment of KTRs to a clinical trial of finerenone with embedded kidney biopsy study. Finerenone is postulated to decrease the risk of kidney and cardiovascular events in KTRs, unrelated to the immunologic inciting factors or mediators of acute rejection episodes. In essence, it is hypothesized that the mechanisms by which finerenone decreases kidney and cardiovascular endpoints in people with type 2 diabetes (T2D) and native CKD, will be similarly effective in patients (regardless of diabetes status) living with a kidney transplant. It is unknown to what extent KTRs and their treating transplant physicians would be willing to participate in a clinical trial of a drug that is targeted at 'general' reduction of CKD and cardiovascular outcomes. In particular, this trial could help provide strategies for successful recruitment of KTRs into such trials.

Kidney tissue is a particularly valuable tool for identifying mechanisms through which finerenone may decrease progression of interstitial fibrosis and CNIT in KTRs. Such information is deemed critical in helping to determine whether future, larger trials of KTRs are indicated, and whether kidney biopsy could be useful for stratifying participants (eg. based on the presence or degree of interstitial fibrosis). Kidney biopsy also yields valuable information helpful to clinical decisions in caring for KTRs but does come with some risks. Thus, the feasibility of enrolling KTRs to a 'not for cause' kidney biopsies in the context of a clinical trial targeting CKD and Cardiovascular Disease (CVD) is unknown.

Objective 2: To measure the tolerability and safety of finerenone in KTRs. Finerenone has not been administered in KTRs and it is unclear whether tolerability will be similar to that of people with diabetes (and perhaps those without) and CKD. The primary concerns include risks for hyperkalemia and creatinine fluctuations which may necessitate temporary or permanent withdrawal of finerenone and also result in downstream interventions specific to kidney transplantation. Immunosuppression for KTRs most often includes a calcineurin inhibitor (CNI) which increases the risk for hyperkalemia, as does finerenone. Moreover, many KTRs are also treated with renin angiotensin system (RAS) blockers, which only further increases this risk. This study will help determine the magnitude of this risk, optimal approaches to managing hyperkalemia specifically in KTRs, and which subpopulations are less likely to tolerate finerenone (eg. those on CNI and RAS blockers), in order to inform potential future clinical trials. The other concern for tolerability of finerenone in KTRs, is the tendency in clinical practice to discontinue medications with the potential to reduce eGFR in KTRs when creatinine levels rise, in order to assess whether rejection is in progress. Ultimately, if KTRs are not able to be maintained on finerenone for a reasonable period, it is unlikely that they would experience potential benefits either. Tolerability will be measured by the relative time on study drug in the two comparator groups.

Safety analyses will build further upon the outcomes of tolerability and will include: hyperkalemia (>5.5m Eq/L), other hyperkalemia-associated events designated by the investigator as requiring holding/discontinuing study drug or RAS blocker, and acute kidney injury episodes defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria, infections requiring acute care (emergency room visits or hospitalization).

Objective 3: To determine the effect of finerenone on clinical, radiologic and pathologic kidney markers in KTRs. Finerenone decreases the risk for progression of CKD and CV events in people with T2D and CKD. It is likely that the effect is similar, regardless of diabetes status, and trials are underway to determine this. KTRs have several potential confounding factors relating to the pathogenesis of worsening kidney disease, namely use of CNIs, donor derived disease, BK virus associated nephropathy and other urinary tract infections, and both acute and chronic T cell or antibody mediated rejection, which may override any potential benefit from finerenone. Alternatively, the anti-inflammatory and antifibrotic effects of finerenone may be particularly beneficial in KTRs with chronic kidney dysfunction secondary to any of the above processes as the final common pathway that results in allograft dysfunction and failure in all of the above is inflammation and fibrosis.

CV disease is a major burden in KTRs, with event rates higher than in the general population, which may partly be related to the fact that most KTRs spend several years on dialysis prior to transplantation. KTRs are at also at high risk of other complicating/competing factors linked to CV events, including the vascular impact of immunosuppressive agents, infection and malignancy. It is unknown whether the complex health status and treatments of KTRs will alter the potential benefit of finerenone on CV events and death.

This relatively short-term trial will include multiple exploratory clinical, radiologic and pathologic endpoints. Exploratory clinical kidney and CV endpoints will focus on relative changes in albuminuria, eGFR slope and the relative difference in the need for acute care for congestive heart failure. Exploratory radiologic endpoints include kidney cortical perfusion, oxygenation and fibrosis as measured by fMRI, and pathologic parameters are to include changes in Banff classification, percent change in interstitial fibrosis using sirius red staining. Blood, urine and kidney specific cytokines and fibrotic markers will also be measured at baseline and at the end of active treatment.

ELIGIBILITY:
Clinical Trial Inclusion Criteria:

* Adult kidney transplant recipients ≥ 18 years
* 1 to 10 years post kidney transplantation from a deceased or living donor
* Stable kidney allograft function (within 20% baseline eGFR) and based on the clinical judgement of the investigator
* Preserved kidney allograft function defined as an eGFR ≥ 25 mL/min/1.73 m
* Urine albumin:creatinine ratio (UACR) ≥30 ug/mg
* Ability of the participant, or their legally authorized representative, to provide informed consent
* Contraceptive requirements:
* Women of non-childbearing potential do not need to undergo pregnancy testing or agree to use adequate contraception. Non-childbearing potential is defined as documented hysterectomy, bilateral salpingectomy, oophorectomy or postmenopausal females (amenorrhea for 12 months without an alternative medical cause). A single high follicle stimulating hormone level in the postmenopausal range may be used to confirm a postmenopausal state.
* Women of childbearing potential can only be included if a pregnancy test is negative at the screening visit and if they agree to use adequate contraception during the study and until 8 weeks after the last study intervention dose. Adequate contraception is defined as an intrauterine device, implant or combined oral contraceptive with a physical barrier (e,g., condom).

Additional Inclusion Criteria for Kidney Biopsy Sub-study:

* Willingness to undergo research study biopsies at screening and following the 12 month treatment period
* Ability to safely discontinue antiplatelet or anticoagulant treatments
* No known intrinsic bleeding diathesis
* Hemoglobin >9.0 g/dL; Platelets > 100,000; International Normalised Ratio (INR) <1.4 on the day of kidney biopsy
* Body mass index <40
* Blood pressure controlled on the day of biopsy to <160/90

Medical Condition Exclusion Criteria:

* Documented recurrent lupus nephritis, ANtineutrophilic Cytoplasmic Antibody (ANCA) vasculitis, membranoproliferative glomerulonephritis (including C3 glomerulopathy)
* History of solid organ transplantation other than kidney
* Acute kidney injury requiring dialysis within 6 months prior to screening
* Uncontrolled hypertension with a sitting Systolic Blood Pressure (SBP) ≥180 mmHg or Diastolic Blood Pressure (DBP) ≥100 mmHg
* Any indication for treatment with a steroidal MRA
* UACR >3500 mg/g at screening. This may be reassessed if one of the three first morning urine samples is >3500 mg/g at the screening visit
* CV event within 3 months prior to screening (heart failure requiring acute care, myocardial infarction, stroke, transient ischemic attack, pulmonary embolism, elective coronary artery bypass grafting)
* Elective percutaneous coronary intervention within 1 month prior to screening
* Known hypersensitivity to the study treatment
* Addison's disease
* Hepatic insufficiency classified as Child-Pugh C
* Pregnancy, breast feeding or intention to become pregnant

Concomitant Therapies Exclusion Criteria:

* Concomitant therapy with spironolactone, eplerenone, sacubitril/valsartan combination, or potassium-sparing diuretic which cannot be discontinued at least 2 weeks prior to screening
* Simultaneous use of Angiotensin-Converting Enzyme Inhibitors (ACEI) and Angiotensin Receptor Blockers (ARB), without being able to discontinue one of these at least 2 weeks prior to screening
* Use of potent CYP3A4 inhibitors or inducers (to be stopped at least 7 days before randomization).

Other Exclusion Criteria:

* Participation in the MRI Study is excluded for certain pacemakers, electronic implants, shrapnel of the eye and certain types of aneurysm clips.
* Any other history, condition, or therapy which could, in the opinion of the investigator, affect compliance with the study treatment and procedures
* Close affiliation with the investigational site, investigators or staff
* Simultaneous participation in another interventional trial within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment to the main clinical trial: Total number of participants who were eligible and enrolled in the main clinical trial | Up to 3 months after launching the full study protocol
  Signed consent by 30 participants for the main clinical trial within 3 months of launching the full study protocol (date of first person randomized).
Feasibility of recruitment to the kidney biopsy substudy: Total number of participants who were eligible and enrolled in the kidney biopsy substudy | Up to 3 months after launching the full study protocol
  Signed consent by 10 participants for the biopsy substudy within 3 months of launching the full study protocol (date of first person randomized).

SECONDARY OUTCOMES:
Relative tolerability of finerenone | From randomization to last on study drug visit, approximately 12 months
  Relative tolerability is defined as the percent time spent on the investigational product.
Risk for discontinuation of finerenone | From randomization to last on study drug visit, approximately 12 months
  The number of the participants who permanently discontinue the investigational product prior to the last on study drug visit, divided by the total number of study participants in the same treatment group.
Overall safety of finerenone | From randomization to last on study drug visit, approximately 12 months
  The percentage of participants suffering a serious adverse event or adverse event of interest (hyperkalemia, acute kidney injuries) while on study drug.
Adverse Event (AE) related to hyperkalemia | From randomization to last on study drug visit, approximately 12 months
  The percentage of participants requiring acute care (hospitalization or ER visit) for hyperkalemia, while on study drug.
Adverse Event (AE) related to acute kidney injury | From randomization to last on study drug visit, approximately 12 months
  The percentage of participants requiring acute care (hospitalization or ER visit) for acute kidney injury while on study drug.
Efficacy for albuminuria reduction | From randomization to last on study drug visit, approximately 12 months
  The relative Urine Albumin Creatinine Ratio (UACR) reduction between groups, with comparison testing using Kruskal Wallis test. The relative reduction in log transformed mean UACR = 1- logUACR(Last on-drug) / logUACR(Screen).
Efficacy for prevention of congestive heart failure (CHF) | From randomization to last on study drug visit, approximately 12 months
  Relative risk of CHF requiring acute care = [total number of persons with an event in finerenone group/total number of participants in finerenone group] divided by the [total number of persons with an event in finerenone group/total number of participants in finerenone group]

OTHER OUTCOMES:
Efficacy for functional Magnetic Resonance Imaging (fMRI) kidney oxygenation | From within 2 weeks before randomization, within 2 weeks before last on study drug visit, up to 12.5 months
  Difference between active versus placebo groups with respect to absolute change in fMRI measures of cortical oxygen availability, estimated by R2* (s-1) using blood oxygenation level dependent (BOLD) MRI
Efficacy for functional Magnetic Resonance Imaging (fMRI) kidney perfusion | From within 2 weeks before randomization, within 2 weeks before last on study drug visit, up to 12.5 months
  Difference between active versus placebo groups with respect to absolute change in fMRI measures of cortical perfusion (ml/min/100g), estimated using arterial spin labeling (ASL) MRI
Efficacy for functional Magnetic Resonance Imaging (fMRI) kidney fibrosis | From within 2 weeks before randomization, within 2 weeks before last on study drug visit, up to 12.5 months
  Difference between active versus placebo groups with respect to absolute change in fMRI cortical fibrosis, estimated by apparent diffusion coefficient (ADC), (x10-3/s) using diffusion-weighted MRI.
Efficacy for interstitial fibrosis and tubular atrophy (IFTA) | From within 2 weeks before randomization, within 2 weeks before last on study drug visit, up to 12.5 months
  Difference between active versus placebo groups with respect to absolute change in percent of cortex with IFTA

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mottl, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Prabir Roy-Chaudhury, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Eastowne Kidney Transplant Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared from 9 through 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 9 months through 36 months after publication
Access Criteria: The investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with University of North Carolina (UNC).

REFERENCES:
- [Background] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Background] Hart A, Lentine KL, Smith JM, Miller JM, Skeans MA, Prentice M, Robinson A, Foutz J, Booker SE, Israni AK, Hirose R, Snyder JJ. OPTN/SRTR 2019 Annual Data Report: Kidney. Am J Transplant. 2021 Feb;21 Suppl 2:21-137. doi: 10.1111/ajt.16502. PMID 33595191
- [Background] Rangaswami J, Mathew RO, Parasuraman R, Tantisattamo E, Lubetzky M, Rao S, Yaqub MS, Birdwell KA, Bennett W, Dalal P, Kapoor R, Lerma EV, Lerman M, McCormick N, Bangalore S, McCullough PA, Dadhania DM. Cardiovascular disease in the kidney transplant recipient: epidemiology, diagnosis and management strategies. Nephrol Dial Transplant. 2019 May 1;34(5):760-773. doi: 10.1093/ndt/gfz053. PMID 30984976
- [Background] Matas AJ, Humar A, Gillingham KJ, Payne WD, Gruessner RW, Kandaswamy R, Dunn DL, Najarian JS, Sutherland DE. Five preventable causes of kidney graft loss in the 1990s: a single-center analysis. Kidney Int. 2002 Aug;62(2):704-14. doi: 10.1046/j.1523-1755.2002.00491.x. PMID 12110036
- [Background] Paraskevas S, Kandaswamy R, Humar A, Gillingham KJ, Gruessner RW, Payne WD, Najarian JS, Sutherland DE, Matas AJ. Risk factors for rising creatinine in renal allografts with 1 and 3 yr survival. Clin Transplant. 2006 Nov-Dec;20(6):667-72. doi: 10.1111/j.1399-0012.2006.00566.x. PMID 17100713
- [Background] Morales JM, Marcen R, del Castillo D, Andres A, Gonzalez-Molina M, Oppenheimer F, Seron D, Gil-Vernet S, Lampreave I, Gainza FJ, Valdes F, Cabello M, Anaya F, Escuin F, Arias M, Pallardo L, Bustamante J. Risk factors for graft loss and mortality after renal transplantation according to recipient age: a prospective multicentre study. Nephrol Dial Transplant. 2012 Dec;27 Suppl 4(Suppl 4):iv39-46. doi: 10.1093/ndt/gfs544. PMID 23258810
- [Background] Karthikeyan V, Karpinski J, Nair RC, Knoll G. The burden of chronic kidney disease in renal transplant recipients. Am J Transplant. 2004 Feb;4(2):262-9. doi: 10.1046/j.1600-6143.2003.00315.x. PMID 14974949
- [Background] Knoll GA. Proteinuria in kidney transplant recipients: prevalence, prognosis, and evidence-based management. Am J Kidney Dis. 2009 Dec;54(6):1131-44. doi: 10.1053/j.ajkd.2009.06.031. Epub 2009 Sep 2. PMID 19726115
- [Background] Lam NN, Tonelli M, Lentine KL, Hemmelgarn B, Ye F, Wen K, Klarenbach S. Albuminuria and posttransplant chronic kidney disease stage predict transplant outcomes. Kidney Int. 2017 Aug;92(2):470-478. doi: 10.1016/j.kint.2017.01.028. Epub 2017 Mar 31. PMID 28366228
- [Background] Gaston RS, Fieberg A, Hunsicker L, Kasiske BL, Leduc R, Cosio FG, Gourishankar S, Grande J, Mannon RB, Rush D, Cecka JM, Connett J, Matas AJ. Late graft failure after kidney transplantation as the consequence of late versus early events. Am J Transplant. 2018 May;18(5):1158-1167. doi: 10.1111/ajt.14590. Epub 2017 Dec 5. PMID 29139625
- [Background] Meier-Kriesche HU, Baliga R, Kaplan B. Decreased renal function is a strong risk factor for cardiovascular death after renal transplantation. Transplantation. 2003 Apr 27;75(8):1291-5. doi: 10.1097/01.TP.0000061602.03327.E2. PMID 12717218
- [Background] Lenihan CR, Liu S, Deswal A, Montez-Rath ME, Winkelmayer WC. De Novo Heart Failure After Kidney Transplantation: Trends in Incidence and Outcomes. Am J Kidney Dis. 2018 Aug;72(2):223-233. doi: 10.1053/j.ajkd.2018.01.041. Epub 2018 Mar 29. PMID 29605378
- [Background] Awan AA, Niu J, Pan JS, Erickson KF, Mandayam S, Winkelmayer WC, Navaneethan SD, Ramanathan V. Trends in the Causes of Death among Kidney Transplant Recipients in the United States (1996-2014). Am J Nephrol. 2018;48(6):472-481. doi: 10.1159/000495081. Epub 2018 Nov 23. PMID 30472701
- [Background] Gaston RS, Fieberg A, Helgeson ES, Eversull J, Hunsicker L, Kasiske BL, Leduc R, Rush D, Matas AJ; DeKAF Investigators*. Late Graft Loss After Kidney Transplantation: Is "Death With Function" Really Death With a Functioning Allograft? Transplantation. 2020 Jul;104(7):1483-1490. doi: 10.1097/TP.0000000000002961. PMID 31568212
- [Background] Ying T, Shi B, Kelly PJ, Pilmore H, Clayton PA, Chadban SJ. Death after Kidney Transplantation: An Analysis by Era and Time Post-Transplant. J Am Soc Nephrol. 2020 Dec;31(12):2887-2899. doi: 10.1681/ASN.2020050566. Epub 2020 Sep 9. PMID 32908001
- [Derived] Vinson AJ, Matas A. Late Allograft Loss and Contemporary Cardiorenal Metabolic Therapies. J Am Soc Nephrol. 2025 Apr 7;36(8):1659-1667. doi: 10.1681/ASN.0000000726. PMID 40193211
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- See also: USRDS Annual Data Report 2020 — https://usrds-adr.niddk.nih.gov/2020
- See also: Organ Procurement and Transplantation Network — https://optn.transplant.hrsa.gov/data/view-data-reports/national-data/